CLINICAL TRIAL: NCT05003609
Title: A Randomised Controlled Trial of Early Rehabilitation in Patients on Extracorporeal Membrane Oxygenation (ECMO-Rehab)
Brief Title: Early Rehabilitation in Patients on Extracorporeal Membrane Oxygenation
Acronym: ECMO-Rehab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Monash University (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANZIC-RC/ECMO-REHAB/001
Record Dates: First submitted 2021-07-14; First posted 2021-08-12 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: Rehabilitation; ECMO

STUDY DESIGN:
Intervention Model Description: 1;1 allocation, stratified by site,
Who Masked: Outcomes Assessor
Masking Description: Blinded outcome assessor - blinded / different therapist (strength) and central follow-up for blinded assessment of PROMs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): ECMO early rehabilitation is led by a senior physiotherapist who has specialised training in ECMO care and coordinates individualised early physical training from randomisation to day 28 in ICU and liaises with the patient through to hospital discharge. The early rehabilitation intervention involves physical activity, functional retraining, strengthening exercises and mobilisation based on a reproducible, physiological approach.
  Interventions: Other: Early Rehabilitation
- Control Group (No Intervention): The control group will receive standard care from nursing and physiotherapy staff not involved in the early, co-ordinated rehabilitation.

INTERVENTIONS:
Other: Early Rehabilitation — The intervention involves a progression of rehabilitation exercises with the objective of rehabilitating the patient at the highest level of exercise possible for the patient for the longest period of time that can be tolerated (up to 60 mins) at each session. The intervention will be administered 5 days per week (weekdays) while the patient remains in ICU, censored at 28 days after randomisation.
  Arms: Intervention Group

SUMMARY:
Critically ill patients who require extracorporeal membrane oxygenation (ECMO) are the sickest in the hospital. More patients are surviving but survivors have compromised functional recovery for months or years. This registry-embedded randomised trial aims to determine if early rehabilitation commenced within 72 hours of ECMO is feasible and improves muscle strength and functional status in patients compared to standard practice in a randomised controlled trial of 100 ICU patients. The effect of the intervention on mortality, health status, and function at 180 days will be evaluated, as well as cost-effectiveness. ECMO-Rehab trial is a registry embedded trial and will be utilising EXCEL data.

DETAILED DESCRIPTION:
The trial is a 100-patient, multicentre, randomised, controlled, parallel-group, two-sided superiority trial that will randomly allocate eligible patients to early rehabilitation or standard care in a 1:1 ratio to determine if early rehabilitation of critically ill patients receiving ECMO reduces disability when compared with standard care. ECMO-Rehab trial is a registry embedded trial and will be utilising EXCEL data.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is on ECMO and expected to remain on ECMO for at least 24 hours
2. Patient is aged 18 years or older.
3. Patient was functionally independent prior to the current admission.
4. Patient is eligible for Medicare (Australian sites only).

Exclusion Criteria:

1. Patient has been receiving ECMO for more than 72 hours.
2. Patient has been in ICU for more than 5 days.
3. Patient has suspected or proven primary myopathic or neurological process associated with prolonged weakness or acute brain injury.
4. Death is deemed imminent by the treating clinician.
5. Patient has a documented medical diagnosis of cognitive impairment e.g. dementia.
6. Patient was unable to mobilise prior to this admission.
7. Patient is unable to communicate in local language.
8. Patient is known to be pregnant.
9. Patient is unlikely to be contactable for 6 months follow-up, e.g. overseas resident, incarcerated
10. The treating clinician does not believe it is in the best interests of the patient to participate in the study
11. Patient who has a bidirectional cannula in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 180 days post randomisation
  The Modified Rankin Scale (mRS) is a 7-level ordered categorical scale capturing levels of patient disability and dependence, with scores ranging from 0 (no disability) to 6 (dead).

SECONDARY OUTCOMES:
Muscle strength at day 14 (Medical Research Council Sum-Score) | 14 days post randomisation
  Grade 0 to Grade 5 where Grade 5 is the best outcome
ECMO-free days to day 28 | 28 days post randomisation
Organ failure free days to day 28 | 28 days post randomisation
Delirium-free days to day 28 | 28 days post randomisation
Activities of Daily Living (ADL) at hospital discharge | up to day of hospital discharge, an average of 3 months
Length of stay on ECMO, in ICU and in hospital | up to day of stay on ECMO, ICU and hospital, an average of 3 months
Mortality rate at ICU and hospital discharge, day 90 and day 180 | up to 180 days post randomisation
Instrumental activities of daily living at 180 days | 180 days post randomisation
  Physical function measured with instrumental activities of daily living
Montreal Cognitive Assessment (MoCA-Blind) | 180 days post randomisation
  Rapid screening instrument for mild cognitive dysfunction. Normal is equal or more than 18 points.
WHO Disability Assessment Schedule 2.0 at day 180 | 180 days post randomisation
  Scoring 10-48 are likely to have clinically significant disability.
Health related quality of life (EQ5D-5L) at day 180 | 180 days post randomisation
  Level of severity 1 to 5 where 5 is the most severe
Daily longitudinal ordinal organ support outcome to day 28 | 28 days post randomisation
  This includes outcomes on Dead; on ECMO; Off ECMO on IMV; Off IMV, in ICU; On acute hospital ward; Discharged alive
Healthcare costs at day 180 | 180 days post randomisation
  Index hospital admission costs will be determined using clinical costing systems at each participating site. Post discharge costs will be determined using patient-level data linkage to determine long-term health care use (including readmission to hospital).
Cost-effectiveness at day 180 | 180 days post randomisation
  The primary cost-effectiveness analysis will be conducted from the Australian healthcare payer's perspective using an analytical time horizon of 180 days.

OTHER OUTCOMES:
Incidence of adverse events | Up to 28 days post randomisation
  Number of patients who suffered adverse events and serious adverse events such as fall, heart attack or new or increased oozing around cannulae during rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, Principal Investigator — ANZIC-RC, Monash University
Locations (7):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Alfred Health, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Toronto General Hospital, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ECMO-PT Study Investigators; International ECMO Network. Early mobilisation during extracorporeal membrane oxygenation was safe and feasible: a pilot randomised controlled trial. Intensive Care Med. 2020 May;46(5):1057-1059. doi: 10.1007/s00134-020-05994-8. Epub 2020 Mar 16. No abstract available. PMID 32179935